CLINICAL TRIAL: NCT00832052
Title: An Investigator And Subject-Blind Phase 1 Study To Characterize The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Doses Of PF-04447943 Up To An Exposure Cap In Healthy Elderly Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, Plasma Drug Levels, and Cognitive Response Following Multiple Doses of a Drug in Healthy Elderly Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0401009
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Healthy; Elderly
Keywords: elderly, multi-dose, safety, efficacy
MeSH Terms: interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Subjects will be randomized to receive either experimental drug (n=6) or placebo (n=2).
  Interventions: Drug: PF-04447943
- Cohort 2 (Experimental): Subjects will be randomized to receive either experimental drug (n=6) or placebo (n=2).
  Interventions: Drug: PF-04447943
- Cohort 3a (Experimental): Subjects will be randomized to receive either experimental drug (n=3) or placebo (n=1).
  Interventions: Drug: PF-04447943
- Cohort 3b (Experimental): Subjects will be randomized to receive either experimental drug (n=3) or placebo (n=1).
  Interventions: Drug: PF-04447943
- Cohort 4 (Experimental)
  Interventions: Drug: PF-04447943

INTERVENTIONS:
Drug: PF-04447943 — Planned oral dose is PF-04447943, 5 mg q12 hours for 7 days.
  Arms: Cohort 1
Drug: PF-04447943 — Planned oral dose is PF-04447943, 15 mg q12 hours for 7 days.
  Arms: Cohort 2
Drug: PF-04447943 — Planned oral dose is PF-04447943, 35 mg q12 hours for 7 days. Actual dose may be adjusted based on pharmacokinetic and other data from prior dose cohorts.
  Arms: Cohort 3a
Drug: PF-04447943 — Planned oral dose is PF-04447943, 35 mg q12 hours for 7 days. Actual dose may be adjusted based on pharmacokinetic and other data from prior dose cohorts.
  Arms: Cohort 3b
Drug: PF-04447943 — Planned oral dose is PF-04447943, 35 mg q12 hours for 14 days. Actual dose may be adjusted downward based on pharmacokinetic and other data from prior dose cohorts.
  Arms: Cohort 4

SUMMARY:
Evaluate the safety and tolerability of PF-04447943 after administration of multiple doses in healthy elderly participants. Evaluate plasma drug levels and effects on cognition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects.
* Subjects must be in reasonably good health as determined by the investigator based on medical history, full physical examination (including blood pressure and pulse rate measurement), 12 lead ECG and clinical laboratory tests.
* Subjects with mild, chronic, stable disease (eg, controlled hypertension, non-insulin dependent diabetes, osteoarthritis may be enrolled if deemed medically prudent by the investigator.
* Subjects taking daily prescription or non-prescription medications for management of acceptable chronic medical conditions must be on a stable dose.
* Body Mass Index (BMI) between 18 to 30 kg/m2, inclusive; and a total body weight >50 kg (110 lbs).
* Creatinine clearance greater than 30 mL/min using the Cockcroft-Gault method.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, immunologic, or allergic disease.
* Use of tobacco or any form of nicotine in the past 6 months.
* Greater than 7 drinks of alcohol per week for women, and greater than 14 drinks of alcohol per week for men.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety endpoints include evaluation of adverse events, change from baseline in vital signs, triplicate and single ECGs, and clinical safety laboratory tests | For cohorts 1-3, up to 17 days; for cohort 4, up to 24 days.
Pharmacokinetic endpoints include plasma PF-04447943 area udner the curve (AUCt ), maximum plasma concentration (Cmax) and time of maximum plasma concentration (Tmax) | For cohorts 1-3, days 1 and 7; for cohort 4, days 1 and 14
Maximum plasma concentration (Cmax) | 1 hour post dose day 4
Minimum plasma concentration ((Ctrough) | For cohorts 1-3, days 2, 3, 4, and 7; for cohort 4, days 2, 3, 4, 12, and 13
Fraction of the total dose excreted in urine (Fe) and the renal clearance (CLR), and, if the data permit, half-life and the observed exposure accumulation ratio (Ro), and fluctuation index (Cmax: Cmin ratio) following multiple doses | For cohorts 1-3, day 7; for cohort 4, day 14

SECONDARY OUTCOMES:
CogState Phase 1 Battery, to include Detect, Identify, One-Card Learning, Groton Maza Learning, Continuous Paired Associated Learning Test, and Composite Cognitive Score | For cohorts 1-3, up to 17 days; for cohort 4, up to 24 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Gainesville, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401009&StudyName=A%20Study%20to%20Evaluate%20Safety%2C%20Tolerability%2C%20Plasma%20Drug%20Levels%2C%20and%20Cognitive%20Response%20Following%20Multiple%20Doses%20of%20a%20Drug%20in%20Healthy